CLINICAL TRIAL: NCT04298775
Title: Postoperative Urinary Retention in Orthopedic Patients Submitted to Intrathecal Anesthesia With Morphine Versus Intrathecal Anesthesia Without Opioid Associated With Peripheral Nerve Block: a Randomized Clinical Trial
Brief Title: Postoperative Urinary Retention in Orthopedic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20160443
Record Dates: First submitted 2020-02-14; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Urinary Retention; Anesthesia, Spinal; Orthopedic Procedures; Nerve Block
MeSH Terms: conditions — Urinary Retention | interventions — Anesthesia, Spinal; Morphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinal anesthesia with morphine (Active Comparator): This patients received subarachnoid anesthesia with 20 mg of Hyperbaric Bupivacaine + 200 mcg of Morphine
  Interventions: Procedure: spinal anesthesia with morphine
- spinal anesthesia without morphine + peripheral nerve block (Active Comparator): This patients received subarachnoid anesthesia with 20 mg of Hyperbaric Bupivacaine and peripheral nerve block with 0.2 to 0.375% Ropivacaine, in a volume of 20 to 30 mL.
  Interventions: Procedure: spinal anesthesia without morphine + peripheral nerve block

INTERVENTIONS:
Procedure: spinal anesthesia with morphine
  Arms: spinal anesthesia with morphine
Procedure: spinal anesthesia without morphine + peripheral nerve block
  Arms: spinal anesthesia without morphine + peripheral nerve block

SUMMARY:
The objective of this study is to compare the incidence of postoperative urinary retention related to spinal anesthesia with morphine and spinal anesthesia associated with peripheral blockade in orthopedic procedures of lower limbs. Secondary objectives are assessing the incidence of nausea and vomiting; postoperative pain and opioid consumption at 24 hours after surgery with each of the techniques. A total of 52 patients submitted to a lower limb orthopedic procedure were randomized to the intervention groups: spinal anesthesia with morphine versus spinal anesthesia without opioid associated with peripheral nerve block. After surgery, bladder ultrasound will be performed in post-anesthesia care unit to identify urinary retention and patients will be followed for 24 hours to assess outcomes.

DETAILED DESCRIPTION:
This is a randomized clinical trial with simple blinding (the outcome evaluator is blind). Approved by the Ethics and Research Committee of Hospital de Clínicas de Porto Alegre under number 20160043 and Plataforma Brasil CAAE 57623815.1.0000.5327.To calculate the sample size, the program WinPEPI, version 11.43, was used. Considering 80% power, 5% significance level and data reported by Tomaszewski, Balkota and Machowicz (RUPO incidence of 42.86% of the spinal anesthesia group with morphine requiring urinary catheterization and 6.25% in patients undergoing peripheral nerve block ). The sample size found was 26 subjects in each group.

Statistical analysis was performed using SPSS STATISTICS software version 23. Absolute and percentage frequencies were calculated for qualitative variables. And mean, standard deviation and interquartile range for quantitative variables. The normality of the quantitative variables was assessed by the Shapiro-Wilk test. The chi-square test was used to assess the difference in the incidence of catheterization in the two groups and the incidence of nausea and vomiting in 24 hours. To evaluate the difference in the mean time to urination, even after sounding, the Student's t test for independent samples was used. Doses of codeine and morphine at 24 hours and assessment of pain on movement and rest at 12 and 24 hours (by the visual analog scale of pain) were assessed by the Mann Whitney test.

P <0.05 was considered statistically significant. The 52 patients included in the survey were allocated randomly to one of the study groups. Randomization was performed immediately before the interventions studied using the electronic random allocation application Randomizer for Clinical Trial for iPad / iPhone, developed by the company Medsharing (http://www.ecrfmedsharing.com/iphone_ipad_randomization.php).

All patients received spinal anesthesia. The technique included sterile preparation of the puncture site at the L3-L4 or L4-L5 level using Whitacre 27G or 25G needles. Group 1 patients received subarachnoid block with 20 mg of hyperbaric bupivacaine + 200 mcg of morphine and group 2 patients received subarachnoid block with 20 mg of hyperbaric bupivacaine and peripheral nerve block.Peripheral nerve blocks were performed after spinal anesthesia, before the start of the surgical procedure under ultrasound visualization associated with the use of neurostimulator. The choice of the nerve to be blocked was based on the innervation related to analgesia of the surgical site: femoral nerve block or sciatic nerve.

In the post-anesthetic care unit, the following parameters were assessed:

* Need for bladder catheterization;
* Time for spontaneous urination (time in minutes between subarachnoid block and spontaneous urination);
* Presence of pain and the need to use opioids;
* Presence of nausea / vomiting and the need to use antiemetics.

Patients were evaluated at 12 and 24 hours after the surgical procedure for:

* Need for bladder catheterization;
* Time for the first spontaneous urination (with or without previous relief bladder catheter);
* Presence of nausea / vomiting;
* Pain assessment by analogue-visual scale from 0 to 10, at the operated site, at rest and during movement;
* Need to use opioids, noting which opioid and dose used.

The postoperative prescription was standardized:

* Paracetamol 500 mg orally 6/6 hours fixed;
* Dipyrone 1 g intravenous 6/6 hours fixed;
* Codeine 30 mg orally 6/6 hours, if mild to moderate pain using an analogue-visual scale (1 to 6);
* Morphine 3 mg intravenously up to 3/3 hours, if severe pain by analogue-visual scale (7 to 10);
* Ondasentron 4 mg intravenously up to 8/8 hours, if nausea / vomiting is present.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective orthopedic surgeries of the lower limbs
* Possibility and acceptance of performing the surgical procedure under spinal anesthesia
* Minimum hospital stay of 24 hours
* Acceptance and signature of the informed consent form

Exclusion Criteria:

* Subjects who did not understand the Portuguese language
* Patients who did not agree with the informed consent term and / or did not sign
* Patients with a history of urological problems
* Severe cognitive disorders
* Patients who were unable to urinate spontaneously before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-07-13 (Actual); Study Completion 2019-07-13 (Actual)

PRIMARY OUTCOMES:
Postoperative urinary retention | In 24 hours after surgical procedure
  Need for bladder catheterization in the first 24 hours after surgical procedure
Postoperative urinary retention | In 24 hours after surgical procedure
  Time required for first spontaneous urination in the first 24 hours after surgical procedure

SECONDARY OUTCOMES:
Nausea and vomiting | In 24 hours after surgical procedure
  Assess the incidence of nausea and vomiting in the groups studied
Postoperative pain: Visual Analog Scale (VAS) | In 12 and 24 hours after surgical procedure
  Evaluate postoperative pain 12 and 24 hours after the surgical procedure, at rest and on movement. Postoperative pain assessment will be performed using the Visual Analog Scale: Scale from Zero to 10 ( being Zero: without pain and 10: worst pain ever felt)
Opioid consumption | In the first 24 hours after surgical procedure
  Assess morphine and codeine consumption. Dose used in the first 24 hours after surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Carolina L Schiavo, M.D, M.Sc, Principal Investigator — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided